CLINICAL TRIAL: NCT03746353
Title: Early Closure of the Derivative Ileostomy Versus Conventional Closure in Postoperative Patients With Low Anterior Resection for Rectal Cancer
Brief Title: Early Closure Versus Conventional Closure in Postoperative Patients With Low Anteriresection for Rectal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C190-10300-120
Record Dates: First submitted 2018-07-31; First posted 2018-11-19 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Colonic Neoplasms; Ileostomy - Stoma; Colorectal Surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early closure of ileostomy (Experimental): Early clousure of ileostomy before 30 days
  Interventions: Procedure: early ileostomy closure
- Conventional closure of ileostomy (Active Comparator): Conventional closure of ileostomy after 30 days
  Interventions: Procedure: early ileostomy closure

INTERVENTIONS:
Procedure: early ileostomy closure — Assigned interventions Conventional closure of ileostomy: Surgical closure of the protective ileostomy 90 or more days after the proctectomy surgery

SUMMARY:
Colorectal cancer worldwide is the third most common in men and the second in female, although mortality is not as high as its incidence, there is less survival in developing countries. According to data from the World Health Organization, in 2012, there were an estimated 1.4 million cases and 693,900 deaths from this disease. Patients with rectal cancer are frequently taken to resection surgery as a curative management of their malignant pathology, according to the type of resection or reconstruction. In a high number of cases, they are management with colorectal anastomosis with a derivative ileostomy in the same procedure. The closure of this ileostomy is usually done after two to three months of the procedure, however in our environment it could take up to six or twelve months, during which time the patient is exposed to social difficulties, management problems and complications, derived from it. The early closure (7-12 days of its creation) of an ileostomy, despite the little evidence, seems to be a safe, feasible procedure that would save the patient having to live temporarily with an ileostomy.

DETAILED DESCRIPTION:
General purpose:

To compare the frequency of perioperative complications and quality of life between early closure of the derivative ileostomy versus conventional closure in postoperative patients with low anterior resection for rectal cancer.

Materials and methods:

Controlled clinical trial, randomized, to be carried out at the National Cancer Institute of Colombia E.S.E. Eligible candidates for the study will be patients older than 18 years who have undergone a previous resection of the rectum plus a derivative ileostomy for colorectal cancer. All patients eligible for inclusion will undergo computed axial tomography with rectal contrast medium on postoperative day 5. Those who meet the inclusion criteria and do not present any of the exclusion criteria will enter the study, prior willingness to participate by part of the patient and obtaining verbal and written informed consent. Through computer-generated randomization, patients will undergo early closure (between 7 and 12 days after the ileostomy) versus conventional closure (after 90 days or more time from the creation of the ileostomy). A sample size of 81 patients was calculated for each arm. The follow-up will be done in both groups at 3, 6, 9 and 12 months after the creation of the ileostomy, including complications using the Clavien-Dindo classification and quality of life using the FACIT-C format. The statistical analysis will be done by protocol and intention to treat. The perioperative complications associated with the closure of the ileostomy, the complications associated with the presence of ileostomy, hospital stay, and quality of life will be analyzed.

Expected impact:

The investigators hope to find that the early closure of ileostomy in patients during the immediate postoperative period of previous resection due to rectal cancer is safe in terms of morbidity and mortality, feasible and with benefits in quality of life during the immediate postoperative period compared with patients to whom they are closed late (after 3 months).

ELIGIBILITY:
Inclusion criteria:

Patients older than 18 years Diagnosis of Rectal cancer treated at the National Institute of Cancerology and any of the institutions attached to the study

Exclusion criteria:

Complications derived from the anterior resection of the rectum:

* Unresolved intestinal obstruction
* Sepsis
* Organ or space type operative site infection
* Hemodynamic inestability
* Need for reinterventions due to complications
* Coagulopathy
* Active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
perioperative complications | 6 yr
  To compare the frequency of perioperative complications and quality of life between early ( closure of the derivative ileostomy versus conventional closure in postoperative patients with low anterior resection for rectal cancer.
  Using the Clavien-Dindo classification (It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The introduction of the subclasses a and b allows a contraction of the classification into 5 grades (I, II, III, IV and V) depending on the size of the population observed or the of the focus of a study.
  Complications that have the potential for long-lasting disability after patient's discharge (e.g.: paralysis of a voice cord after thyroid surgery) are highlighted in the present classification by a suffix ("d" for disability). This suffix indicates that a follow-up is required to comprehensively evaluate the outcome and related long-term quality of life)

SECONDARY OUTCOMES:
The follow-up for describe complications | 6 yr
  Using the Clavien-Dindo classification (It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The introduction of the subclasses a and b allows a contraction of the classification into 5 grades (I, II, III, IV and V) depending on the size of the population observed or the of the focus of a study.
  Complications that have the potential for long-lasting disability after patient's discharge (e.g.: paralysis of a voice cord after thyroid surgery) are highlighted in the present classification by a suffix ("d" for disability). This suffix indicates that a follow-up is required to comprehensively evaluate the outcome and related long-term quality of life)
Measure quality of life | 6 yr
  Using the FACIT-C format (Version 4)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Carreño, Md, Study Director — Instituto Nacional de Cancerologia, Columbia
Locations (3):
- Colombia (3):
  - Instituto Nacional de Cancerología, Bogota, Cundinamarca
  - Clinica Vida, Medellín
  - Hospital Pablo Tobón Uribe, Medellín

IPD SHARING:
Plan to Share IPD: Undecided